CLINICAL TRIAL: NCT04413487
Title: Strain Echocardiogram in Early Detection of Left Ventricular Dysfunction in Cancer Patients Receiving Chemotherapy
Brief Title: Early Detection of Heart Problems in Cancer Patients Receiving Chemotherapy
Status: Withdrawn | Type: Observational
Why Stopped: Study never started due to change in standard of care guideline
Sponsor: The Guthrie Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 20
Record Dates: First submitted 2019-12-09; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Extra echocardiogram — Subjects will receive an extra echocardiogram after 2 cycles of chemotherapy

SUMMARY:
Subjects will include patients diagnosed with breast cancer or hematological cancer who are planned for chemotherapy treatment with anthracycline or trastuzumab; and who have one or more risk factors for cardiovascular disease. Subjects will received an extra echocardiogram to determine if heart problems can be detected earlier.

DETAILED DESCRIPTION:
* Patients scheduled for potentially cardiotoxic chemotherapy would receive a baseline echocardiogram as per standard protocol which should be covered by the routine insurance
* Follow-up with an extra echocardiogram for research purposes would be performed after 2 cycles of that chemotherapy - supplied by the study
* Clinical assessment at 3 to 6 months including repeat echocardiography as per standard care with the research question as whether any differences in strain pattern between pre-chemo and post 2 cycles studies all identify patients who are more likely to have cardiac issues later.
* Patients will have standard of care visits at 3 month, 6 month and 12 month and will be evaluated for cardiac status and survival.
* Patient records will be reviewed at 5 years to check cardiac status and survival.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 years and above
* Willing and able to provide consent
* Able to read
* Patients diagnosed with breast cancer or hematological cancer who are planned for chemotherapy treatment with anthracycline or trastuzumab.
* Patients at increased risk of cardiotoxicity with one or more risk factors for heart disease:

  * LVEF 50-54% by baseline echocardiogram
  * Age ≥ 65
  * BMI ≥ 30 kg/m2
  * Current or prior anti-hypertensive therapy
  * Diagnosis of coronary artery disease (CAD)
  * Diabetes Mellitus
  * Atrial fibrillation/flutter

Exclusion Criteria:

* Children
* Patients who are pregnant
* Only single encounter without follow up
* Cancer diagnosis other than breast or hematological cancer
* Chemotherapy treatment other than anthracycline or trastuzumab
* No prior chemotherapy treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will include patients diagnosed with breast cancer or hematological cancer who are planned for chemotherapy treatment with anthracycline or trastuzumab; and who have one or more risk factors for cardiovascular disease including LVEF 50-54% by baseline echocardiogram; Age ≥ 65; BMI ≥ 30 kg/m2;current or prior anti-hypertensive therapy; diagnosis of coronary artery disease (CAD); Diabetes Mellitus or Atrial fibrillation/flutter.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-03 (Estimated); Primary Completion 2020-05-28 (Actual); Study Completion 2020-05-28 (Actual)

PRIMARY OUTCOMES:
Change in left ventricular ejection fraction (LVEF) | through study completion, an average of 1 year
  a decrease in LVEF of ≥10 percentage points from baseline to a value of < 50% OR a decrease of LVEF by ≥ 5 percentage points from baseline to LVEF <50% for patients who have a baseline LVEF of 50-54%

SECONDARY OUTCOMES:
Survival status | through study completion, an average of 1 year
  alive or deceased
Change in symptoms that may be indicative of heart failure | through study completion, an average of 1 year
  Presence of absence of symptoms
Change in treatment that may be indicative of heart failure | through study completion, an average of 1 year
  Presence or absence of treatment for heart failure
Change in strain echo that may be indicative of heart failure | through study completion, an average of 1 year
  Presence or absence of heart failure by imaging

CONTACTS AND LOCATIONS:
Overall Officials: Philip Lowry, MD, Principal Investigator — The Guthrie Clinic

IPD SHARING:
Plan to Share IPD: No